CLINICAL TRIAL: NCT00554112
Title: Regulation of B-Cell Function & Glucose Tolerance in Older People
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the VA, per Central Office
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: American Diabetes Association (Other)
Responsible Party: Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDA-2-017-07F
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Aging; Glucose Intolerance
Keywords: Exercise Training; Glucose Intolerance; Human Aging; Insulin Secretion
MeSH Terms: conditions — Glucose Intolerance | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Exercise
  Interventions: Behavioral: Exercise
- 2 (Active Comparator): Exercise
  Interventions: Behavioral: Exercise
- 3 (No Intervention): Control

INTERVENTIONS:
Behavioral: Exercise — Exercise
  Arms: 1; 2

SUMMARY:
This VA CDA-2 proposal will test in detail if lifestyle intervention with aerobic exercise training improves the body's production of insulin in older people at risk to develop diabetes.

DETAILED DESCRIPTION:
There is a high prevalence of type 2 diabetes and impaired glucose tolerance (IGT) in the older population. Aging is associated with insulin resistance and impaired insulin secretion, with greater defects in older people with IGT. Beta-cell dysfunction is critical in the progression from normal glucose to tolerance to IGT and to diabetes.

In the Diabetes Prevention Program (DPP), lifestyle intervention with diet and exercise training significantly lowered the rate of progression from IGT to diabetes, and was particularly effective in older people. The mechanisms of lifestyle changes to prevent diabetes and the effects on beta-cell function remain unclear. Exercise is well-known to increase insulin sensitivity, although exercise effects on beta-cell function have not been specifically assessed. In a pilot study supported by local VA funds, one week of aerobic exercise training improved insulin sensitivity as expected, but also improved beta-cell function in sedentary older people with IGT, with no change in body weight/composition, fasting glucose or lipid/inflammatory parameters.

Based on my current VA RCDA project and the pilot study results, this VA CDA-2 proposal will test in detail the novel overall hypothesis that lifestyle intervention with aerobic exercise training leads to improved beta-cell function in human age-related glucose intolerance. The potential mechanisms of the age-associated decline in beta-cell function and whereby exercise training may improve beta-cell function will also be explored. Beta-cell function will be examined in relation to expected improvements in insulin sensitivity, and the effects of exercise will be isolated with weight maintenance and nutritional balance. The time course of exercise effects over three months, the acute and chronic effects of exercise training on beta-cell function, the effects of high vs. low intensity exercise training, and different important components of beta-cell function will be examined. The interaction between exercise training effects on beta-cell function in older people with IGT and potential mediators including free fatty acids (FFA)/FFA composition, intraabdominal fat, adipocytokines, and incretin hormones will be examined.

In light of the striking effectiveness of the DPP lifestyle intervention to prevent diabetes in older people with IGT, the decline in beta-cell function with even normal human aging, and the importance of beta-cell dysfunction in the progression to diabetes, it is of great interest to further define the potential, novel metabolic effects of exercise training on beta-cell function, particularly in the aging population. This project may provide initial steps to further determine the mechanisms whereby lifestyle changes prevent diabetes. This would provide critical information needed to translate research findings into clinical practice in order to prevent diabetes in the aging veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (defined as activity level of no more than occasional short bouts of walking per week), community-dwelling older veterans and non-veterans age 60-80 years. Special recruitment efforts will focus on enrollment of veterans.
* Fasting glucose <126 mg/dl and 2-hr glucose 140-199 mg/dl (IGT) during OGTT.
* BMI 26-36 kg/m2.

Exclusion Criteria:

* Current use of oral anti-diabetic agents, insulin, systemic steroids, beta-blockers, thiazides.
* Abnormal screening exercise stress test: exercise-induced sustained arrhythmia, symptomatic myocardial ischemia, ischemic EKG changes (>2mm ST-T depression in non Q-wave lead) during screening maximum treadmill test.
* Clinically significant cardiac disease defined as congestive heart failure (CHF) requiring pharmacologic therapy or New York Heart Association (NYHA) Class 3 or 4 cardiac status, atrial fibrillation, symptomatic obstructive valvular disease, high-grade AV block, unstable angina, or myocardial infarction within the last 12 months.
* Participation in a physical therapy, exercise or diet program.
* Significant orthopedic or musculoskeletal conditions.
* Clinically significant renal disease and/or serum creatinine > 2.0 mg/dl.
* Hemoglobin <10 g/l.
* Clinically significant liver disease and/or ALT > 2.5 fold the upper limit of normal.
* Clinically significant medical history or physical findings (e.g. chronic lung disease, cancer) detected at the screening assessment.
* Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Exercise effect on beta-cell function at 3 months | 3 months

SECONDARY OUTCOMES:
Exercise effects glucose tolerance, intraabdominal fat, lipids, glycerol, GLP-1, adiponectin, and leptin. | 3 months